CLINICAL TRIAL: NCT00392743
Title: An Open-label, Cross-over Study, to Compare the PET and SPECT Measurement of Antipsychotic-induced D2 Receptor Occupancy, in a Group of Healthy Volunteers and in Another Group of Patients With Schizophrenia and Other Psychotic Disorders
Brief Title: A Study to Compare Two Different Brain Imaging Techniques in Healthy Volunteers and in Schizophrenic Patients
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: TMT108154
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-10

CONDITIONS: Schizophrenia
Keywords: Bolus; 11C-Raclopride; Schizophrenia; 123I-IBZM; SPECT; Receptor Occupancy; PET; MRI; Antipsychotics; Bolus/Infusion
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pet/spect scan
  Interventions: Procedure: pet/spect scan

INTERVENTIONS:
Procedure: pet/spect scan

SUMMARY:
A direct comparison of Positron Emission Tomography (PET) (11C-Raclopride) and Single Photon Emission Computed Tomography (SPECT) (123I-IBZM) D2 RO measurements would allow GSK to gain understanding on the SPECT results obtained with SB773812, and to accurately interpret future D2 RO results from either PET or SPECT studies with new compounds.

ELIGIBILITY:
Inclusion criteria:

* Not pregnant or becoming pregnant during the study.
* No abnormality in clinical examination, clinical laboratory test or ECG.
* Not taking drugs
* Patients with schizophrenia, schizophreniform disorder or schizoaffective disorders.
* Patients with at least 1 month antipsychotic monotherapy with either risperidone, olanzapine or clozapine.
* Healthy volunteers with no neurological or psychiatric illness.

Exclusion criteria:

* Have received other antipsychotic during the last month or neuroleptics during the last year.
* If you have taken part in investigations you should not receive a radiation dose of more than 10 mSv over any 3 year period.
* History of bleeding disorder or are taking medication that affects blood clotting
* History of substance dependence (except nicotine)
* Claustrophobia
* Gross head deformity.
* Unable to lie still in the PET or SPECT camera for 1 hour and a half.
* The presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a methodology study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
PET and SPECT striatal binding potential | at day 1

SECONDARY OUTCOMES:
plasma concentrations at the time of scanning, | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Espluges de Llobregat
  - GSK Investigational Site, Sant Boi de Llobregat